CLINICAL TRIAL: NCT05912959
Title: Efficacy of Adding Photo Biostimulation to Standard Physical Therapy Treatment for Spastic Calf Muscle on Tone, Gross Motor Function, Planter Surface Area, and Quality of Life
Brief Title: Photo Biostimulation and Spasticity in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, principal investigator, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2023-313
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy; Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: parallel model study where 2 groups (experimental and control) will receive specific interventions. then the outcome measures will be assessed at baseline, after treatment (at 4 weeks) then at 3 month follow up
Who Masked: Participant, Outcomes Assessor
Masking Description: Concealed allocation will be performed by a researcher who will not be involved in the treatment or assessment. Permuted blocks will be used to assure an equal 1:1 allocation ratio. Due to the nature of the study, the assessor and the patients will be blindfolded (double-blinded). During the first treatment session, the therapist will be allowed to uncover the allocation code to be able to conduct the appropriate treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photo biostimulation group (Experimental): * this group will receive a photo bio stimulation (LASER) session consisting of 3 sessions using the LASER device (VECTRA GENISYS, INTELLECT LEGEND XT, Chattanooga, USA). The following parameters will be used; Power output: 300 mv, Wavelength: 820 nm, Contact area: 0.495; Powr density: 0.606 mW/ cm2, Treatment time per point: 13 seconds, Number of points are three: (GB34, LR3, LIV 3).
  * in addition to the LASER, this group will receive a standard physiotherapy program designed by an experienced pediatric physical therapist
  Interventions: Other: photo biostimulation
- standard physiotherapy group (Active Comparator): This group will receive a standard physiotherapy program designed by an experienced pediatric physical therapist
  Interventions: Other: photo biostimulation

INTERVENTIONS:
Other: photo biostimulation — the intervention is a type of wavelength around 820 nm. this method of treatment is totally safe. yet, it has many therapeutic effects on the cellular level as well as tissue and organ level. during treatment with laser, the patient does not feel any specific sensation.
  Other Names: (Low Level Therapeutic LASER); LASER

SUMMARY:
the current study will address the spasticity in calf muscle secondary to cerebral palsy in children. As the spasticity can inversely affect muscle contraction, joint function, and consequently the function and quality of life, the current study will investigate the effect of adding photobiostimulation therapy to standard physiotherapy on muscle tone, ankle range of motion, gross motor function, plantar surface of the affected foot, and quality of life in patients with spastic cerebral palsy

DETAILED DESCRIPTION:
spasticity is one of the common complications associated with upper motor neuron injuries such as cerebral palsy. it can affect the normal developmental process of the child as it restricts muscle performance, limit range of motion, decrease function, and affect the ability to engage in daily activities.

the current study will include 2 groups of children having spastic cerebral palsy. these groups will be randomly distributed to the experimental group (receive standard physiotherapy treatment plus photo biostimulation therapy on related acupuncture points) and the control group will receive a standard physiotherapy program.

the duration of the intervention will be 1 month, 3 sessions per week. the outcome measures will be assessed at baseline, at the end of the intervention ( after 4 weeks of treatment), and at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age between 8 and 14 years,
* who had a diagnosis of spastic cerebral palsy by a pediatrician, with at least one spastic - muscle in the extremities,
* grades 1 -4 on Gross Motor Function Classification System
* score 1 on the Modified Ashworth Scale (MAS)
* the ability to walk alone or with assistance
* whose parents/guardians sign the informed consent form,
* who were willing to complete the study.

Exclusion Criteria:

* patients with anatomical disorders,
* patients who received a botulinum toxin injection in the calf muscle during the last six months
* surgery in the lower extremity during the previous year
* severe associated neurological diseases such as epilepsy
* poor nutritional status,

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth scale for muscle tone assessment | at baseline
  this scale is a simple clinical scale used to assess muscle tone ans spasticity level. it ranges from 1 to 4 where the lowest value indicate normal muscle tone and the largest value indicate high miscle tone
Modified Ashworth scale for muscle tone assessment | after the end of the treatment (after 4 weeks)
  this scale is a simple clinical scale used to assess muscle tone ans spasticity level. it ranges from 1 to 4 where the lowest value indicate normal muscle tone and the largest value indicate high miscle tone
Modified Ashworth scale for muscle tone assessment | at 4 weeks after the end of the treatment (follow-up)
  this scale is a simple clinical scale used to assess muscle tone ans spasticity level. it ranges from 1 to 4 where the lowest value indicate normal muscle tone and the largest value indicate high miscle tone
plantar surface area | at baseline
  A footscan plantar pressure detection system will be used to determine the plantar support area and plantar pressure. This device consists of a force plate (FAS system 1.0 ACP Light, Buratto Advanced Technology, Treviso, Italy), with an active surface (47.5 × 43.0 cm) equipped with 2544 optical sensors distributed along the perimetrical border. it can assess the plantar surface area and the peak pressure in each part of the plantar surface
plantar surface area | at 4 weeks
  A footscan plantar pressure detection system will be used to determine the plantar support area and plantar pressure. This device consists of a force plate (FAS system 1.0 ACP Light, Buratto Advanced Technology, Treviso, Italy), with an active surface (47.5 × 43.0 cm) equipped with 2544 optical sensors distributed along the perimetrical border. it can assess the plantar surface area and the peak pressure in each part of the plantar surface
plantar surface area | at 4 weeks after the end of the treatment (follow-up)
  A footscan plantar pressure detection system will be used to determine the plantar support area and plantar pressure. This device consists of a force plate (FAS system 1.0 ACP Light, Buratto Advanced Technology, Treviso, Italy), with an active surface (47.5 × 43.0 cm) equipped with 2544 optical sensors distributed along the perimetrical border. it can assess the plantar surface area and the peak pressure in each part of the plantar surface
Gross Motor Function Measure (GMFM) (88 items) | at baseline
  Gross Motor Function Measure (GMFM) (88 items) is a tool used to assess changes in gross motor function in cerebral palsy patients. this clinical scale is easy to use and categorize children according to their abilities. where the lower scale mean better gross motor function and higher value means more limitations in gross motor scale
Gross Motor Function Measure (GMFM) (88 items) | at 4 weeks
  Gross Motor Function Measure (GMFM) (88 items) is a tool used to assess changes in gross motor function in cerebral palsy patients. this clinical scale is easy to use and categorize children according to their abilities. where the lower scale mean better gross motor function and higher value means more limitations in gross motor scale
Gross Motor Function Measure (GMFM) (88 items) | at 4 weeks after the end of treatment (follow-up)
  Gross Motor Function Measure (GMFM) (88 items) is a tool used to assess changes in gross motor function in cerebral palsy patients. this clinical scale is easy to use and categorize children according to their abilities. where the lower scale mean better gross motor function and higher value means more limitations in gross motor scale
The pediatric quality of life questionnaire for cerebral palsy | at baseline
  it is a validated tools with strong psychometric properties and clinical utility. The parent proxy's form (parents of children aged 4-12 years) comprises 66 items and the child self-report form (9-12 years) comprises 52 items. Both the child's and the parent proxy's forms have demonstrated good psychometric properties including internal consistency, test-retest reliability, and construct validity. The higher the score, the better the quality of life is represented
The pediatric quality of life questionnaire for cerebral palsy | at 4 weeks
  it is a validated tools with strong psychometric properties and clinical utility. The parent proxy's form (parents of children aged 4-12 years) comprises 66 items and the child self-report form (9-12 years) comprises 52 items. Both the child's and the parent proxy's forms have demonstrated good psychometric properties including internal consistency, test-retest reliability, and construct validity. The higher the score, the better the quality of life is represented
The pediatric quality of life questionnaire for cerebral palsy | at 4 weeks after the end of treatment (follow-up)
  it is a validated tools with strong psychometric properties and clinical utility. The parent proxy's form (parents of children aged 4-12 years) comprises 66 items and the child self-report form (9-12 years) comprises 52 items. Both the child's and the parent proxy's forms have demonstrated good psychometric properties including internal consistency, test-retest reliability, and construct validity. The higher the score, the better the quality of life is represented

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hail, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
this will be discussed with the project funders